CLINICAL TRIAL: NCT02780726
Title: A Phase 3, Multi-center, Open-label Study of Intermittent Oral Dosing of ASP1517 in Peritoneal Dialysis Chronic Kidney Disease Patients With Anemia
Brief Title: A Study of Intermittent Oral Dosing of ASP1517 in Peritoneal Dialysis Chronic Kidney Disease Patients With Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1517-CL-0302
Record Dates: First submitted 2016-05-20; First posted 2016-05-23 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Peritoneal Dialysis Chronic Kidney Disease Patients With Anemia
Keywords: Peritoneal dialysis; Roxadustat; Renal anemia; ASP1517
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASP1517 Low Dose Group (ESA Untreated) (Experimental): This group includes subjects who have not received Erythropoieses Stimulating Agents (ESAs). Study drug will be dosed three times weekly and dose adjustments will be made during the study.
  Interventions: Drug: roxadustat
- ASP1517 High Dose Group (ESA Untreated) (Experimental): This group includes subjects who have not received ESAs. Study drug will be dosed three times weekly and dose adjustments will be made during the study.
  Interventions: Drug: roxadustat
- ASP1517 ESAs Treated Group (Experimental): This group includes subjects who have received ESAs. The treatment was converted from ESAs to study drug. Study drug will be dosed three times weekly and dose adjustments will be made during the study.
  Interventions: Drug: roxadustat

INTERVENTIONS:
Drug: roxadustat — Oral
  Other Names: ASP1517

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of ASP1517 in peritoneal dialysis chronic kidney disease patients with anemia.

ELIGIBILITY:
Inclusion Criteria:

* Female subject must either:

Be of non-childbearing potential:

* post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
* documented surgically sterile Or, if of childbearing potential,
* Agree not to try to become pregnant during the study and for 28 days after the final study drug administration
* And have a negative pregnancy test at Screening
* And, if heterosexually active, agree to consistently use two forms of highly effective form of birth control (at least one of which must be a barrier method) starting at Screening and throughout the study period and continued for 28 days after the final study drug administration.

  * Female subject must agree not to breastfeed starting at Screening and throughout the study period, and continued for 28 days after the final study drug administration.
  * Female subject must not donate ova starting at Screening and throughout the study period, and continued for 28 days after the final study drug administration.
  * Male subject and their female spouse/partners who are of childbearing potential must be using two forms of highly effective form of birth control (at least one of which must be a barrier method) starting at Screening and continue throughout the study period, and for 12 weeks after the final study drug administration
  * Male subject must not donate sperm starting at Screening and throughout the study period and, for 12 weeks after the final study drug administration
  * Subjects who have not received Erythropoieses Stimulating Agents (ESAs):
* Subjects who have been receiving peritoneal dialysis for more than 4 weeks before the screening assessment
* Subjects who have never received ESAs after starting peritoneal dialysis, or subjects who have not received ESAs within 6 weeks before the screening assessment.
* Mean of the subject's two most recent Hb values before randomization during the Screening Period must be <10.5 g/dL with an absolute difference ≤1.3 g/dL between the two values
* Either transferrin saturation (TSAT) ≥ 5% or serum ferritin ≥ 30 ng/mL during the screening period

  * Subjects who have been receiving ESAs:
* Subjects with renal anemia who have been receiving ESA within the doses approved in Japan for more than 8 weeks after starting peritoneal dialysis, before the screening assessment
* Mean of the subject's two most recent Hb values before randomization during the Screening Period must be ≥10.0 g/dL and ≤12.0 g/dL
* TSAT ≥ 20% or serum ferritin ≥ 100 ng/mL during the screening period

Exclusion Criteria:

* Subjects who had trouble with continuing peritoneal dialysis due to peritonitis, development of catheter trouble (e.g. tunnel infection) within 4 weeks before the screening assessment
* Concurrent retinal neovascular lesion requiring treatment and macular edema requiring treatment
* Concurrent autoimmune disease with inflammation that could impact erythropoiesis
* History of gastric/intestinal resection considered influential on the absorption of drugs in the gastrointestinal tract (excluding resection of gastric or colon polyps) or concurrent gastro-paresis
* Uncontrolled hypertension
* Concurrent congestive heart failure (NYHA Class III or higher)
* History of hospitalization for treatment of stroke, myocardial infarction, or pulmonary embolism within 12 weeks before the screening assessment
* Positive for hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (HCV) antibody at the screening assessment, or positive for human immunodeficiency virus (HIV) in a past test
* Concurrent other form of anemia than renal anemia
* Having received treatment with protein anabolic hormone, testosterone enanthate, or mepitiostane within 6 weeks before the screening assessment
* Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), total bilirubin, or Alkaline Phosphatase (ALP) that is greater than the criteria below, or previous or concurrent another serious liver disease at screening assessment
* Previous or current malignant tumor (no recurrence for at least 5 years is eligible.)
* Having undergone blood transfusion and/or a surgical procedure considered to promote anemia (excluding shunt reconstruction surgery for access to the blood) within 4 weeks before the screening assessment
* Having undergone a kidney transplantation
* Having a previous history of treatment with ASP1517
* History of serious drug allergy including anaphylactic shock
* Participation in another clinical study or post-marketing clinical study (including that of a medical device) within 12 weeks before informed consent acquisition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (Hb) Response Rate from Week 18 to Week 24 | Up to Week 24
  Hb response defined as average Hb within the target range in this outcome

SECONDARY OUTCOMES:
Hb Response rate | Up to Week 24
  Hb response is defined as reaching target values for Hb and change of Hb from baseline in this outcome.
Average Hb levels from week 18 to week 24 | Up to week 24
Change from baseline in the average Hb levels of week 18 to week 24 | Baseline and up to Week 24
Rate of rise in Hb levels (g/dL/week) | Up to Week 4
Proportion of time points with target Hb levels | Up to Week 24
Proportion of participants who achieve the target Hb level at each week | Up to Week 24
Proportion of participants who achieve the lower limit of the target Hb level | Up to Week 24
Time to achieve the lower limit of the target Hb level | Up to Week 24
Change from baseline in Hb level at each week | Baseline and Up to Week 24
Efficacy assessed by hematocrit | Up to Week 24
  Hematocrit will be summarized by ASP1517 low dose Erythropoieses Stimulating Agent (ESA) untreated group, ASP1517 high dose ESA untreated group and ASP1517 ESAs treated Group.
Efficacy assessed by reticulocytes/ erythrocytes | Up to Week 24
  Reticulocytes/Erythrocytes will be summarized by ASP1517 low dose ESA untreated group, ASP1517 high dose ESA untreated group and ASP1517 ESAs treated Group.
Efficacy assessed by Iron (Fe) | Up to Week 24
  Fe will be summarized by ASP1517 low dose ESA untreated group, ASP1517 high dose ESA untreated group and ASP1517 ESAs treated Group.
Efficacy assessed by ferritin | Up to Week 24
  Ferritin will be summarized by ASP1517 low dose ESA untreated group, ASP1517 high dose ESA untreated group and ASP1517 ESAs treated Group.
Efficacy assessed by transferrin | Up to Week 24
  Transferrin will be summarized by ASP1517 low dose ESA untreated group, ASP1517 high dose ESA untreated group and ASP1517 ESAs treated Group.
Efficacy assessed by total iron binding capacity | Up to Week 24
  Total iron binding capacity will be summarized by ASP1517 low dose ESA untreated group, ASP1517 high dose ESA untreated group and ASP1517 ESAs treated Group.
Efficacy assessed by soluble transferrin receptor | Up to Week 24
  Soluble transferrin receptor will be summarized by ASP1517 low dose ESA untreated group, ASP1517 high dose ESA untreated group and ASP1517 ESAs treated Group.
Efficacy assessed by transferrin saturation | Up to Week 24
  Transferrin saturation will be summarized by ASP1517 low dose ESA untreated group, ASP1517 high dose ESA untreated group and ASP1517 ESAs treated Group.
Efficacy assessed by reticulocyte hemoglobin content | Up to Week 24
  Reticulocyte hemoglobin content will be summarized by ASP1517 low dose ESA untreated group, ASP1517 high dose ESA untreated group and ASP1517 ESAs treated Group.
Quality of life assessed by SF-36 | Up to Week 24
  SF-36: Medical Outcomes Study 36-Item Short-Form Health Survey
Quality of life assessed by EQ-5D | Up to Week 24
  EQ-5D: EuroQol 5 Dimension
Quality of life assessed by FACT-An | Up to Week 24
  FACT-An: Functional Assessment of Cancer Therapy-Anemia
Occurrence of hospitalizations | Up to Week 24
Safety assessed by incidence of adverse events | Up to Week 24
Number of participants with abnormal Vital signs and/or adverse events related to treatment | Up to Week 24
Safety assessed by standard 12-lead electrocardiogram | Up to Week 24
Number of participants with abnormal Laboratory values and/or adverse events related to treatment | Up to Week 24
Plasma concentration of unchanged ASP1517 | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (15):
- Japan (15):
  - Site JP00002, Aichi
  - Site JP00004, Aichi
  - Site JP00010, Aichi
  - Site JP00013, Aichi
  - Site JP00001, Fukuoka
  - Site JP00005, Fukuoka
  - Site JP00012, Hokkaido
  - Site JP00014, Hokkaido
  - Site JP00006, Ishikawa
  - Site JP00008, Kanagawa
  - Site JP00003, Nagano
  - SIte JP00015, Okayama
  - Site JP00009, Osaka
  - Site JP00007, Tokushima
  - Site JP00011, Toyama

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Hamano T, Yamaguchi Y, Goto K, Mizokawa S, Ito Y, Dellanna F, Barratt J, Akizawa T. Risk Factors for Thromboembolic Events in Patients With Dialysis-Dependent CKD: Pooled Analysis of Phase 3 Roxadustat Trials in Japan. Adv Ther. 2024 Apr;41(4):1526-1552. doi: 10.1007/s12325-023-02727-3. Epub 2024 Feb 16. PMID 38363463
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=354